CLINICAL TRIAL: NCT05681403
Title: Clinical Study of Mitoxantrone Hydrochloride Liposome, Carmostine, Etoposide and Cytarabine as Conditioning Regimen for Autologous Hematopoietic Stem Cell Transplantation in Patients With Lymphoma
Brief Title: Clinical Study of Improved BEAM Conditioning Regimen for ASCT in Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSK-238
Record Dates: First submitted 2022-12-11; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-10

CONDITIONS: Lymphoma; Autologous Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Improved BEAM regimen (Experimental): The enrolled subjects will received mitoxantrone hydrochloride liposome, carmostine, etoposide and cytarabine as conditioning regimen for ASCT.
  Interventions: Drug: Improved BEAM regimen

INTERVENTIONS:
Drug: Improved BEAM regimen — Mitoxantrone hydrochloride liposome, carmostine, etoposide and cytarabine will be used as conditioning regimen for ASCT in the lymphoma patients.
  Other Names: Conditioning treatment with improved BEAM regimen

SUMMARY:
This is a single arm, open, single-center clinical study. The patients who are diagnosed with lymphoma and intend to undergo ASCT will be enrolled. The aim of this study is to investigate the efficacy and safety of the conditioning regimen using mitoxantrone hydrochloride liposome, BCNU, etoposide and cytarabine for ASCT.

DETAILED DESCRIPTION:
High-dose chemotherapy combined with autologous hematopoietic stem cell transplantation (ASCT) is considered the standard of care for patients with chemotherapy-sensitive relapsed/refractory (R/R) non-Hodgkin's lymphoma (NHL). BEAM regimen is the most commonly used conditioning regimen for ASCT in lymphoma. But its application is limited by the adverse drug reactions. This present project is a one-arm, open, single-center clinical study. It aims to evaluate the efficacy and safety of mitoxantrone hydrochloride liposome, carmostine, etoposide, and cytarabine as the conditioning regimen for ASCT in patients with lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Subjects volunteered to join the study, signed informed consent, had good compliance, and cooperated with follow-up.
* Aged 18-60 years, male or female.
* Subjects pathologically diagnosed non-Hodgkin's lymphoma, and intend to undergo autologous hematopoietic stem cell transplantation.
* ECOG score 0-1.
* Meet the following requirements: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 times the upper limit of normal value (ULN), total bilirubin (TBIL) ≤1.5×ULN (AST and ALT≤5×ULN are allowed if liver invasion occurs); serum creatinine ≤1.5×ULN; international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤1.5×ULN; ECG examination was normal or abnormal without clinical significance, cardiac ultrasound showed left ventricular ejection fraction (LVEF) greater than 60, or CK-MB is normal, pro-BNP less than 900 pg/mL.
* Female subjects have negative serum pregnancy test result. Subjects use highly effective birth control methods throughout the trial.

Exclusion Criteria:

* Previous recipients of mitoxantrone or mitoxantrone liposome; previous treatment with doxorubicin or other anthracyclines, with a cumulative dose of doxorubicin > 360 mg/m2 (for other anthracyclines, 1 mg doxorubicin is equivalent to 2 mg epirubicin).
* Hypersensitivity to any study drug or its component.
* Uncontrolled systemic diseases (e.g., active infections, uncontrolled hypertension, diabetes, etc.) .
* Cardiac function and disease meet one of the following conditions: a) Long QTc syndrome or QTc interval >480 ms; b) Complete left bundle branch block, degree II or III atrioventricular block; c) Severe uncontrolled arrhythmias that require medical treatment; d) New York College of Cardiology Grade ≥ III; e) Cardiac ejection fraction (LVEF) less than 60%; f) A history of myocardial infarction, unstable angina pectoris, severely unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities within 6 months prior to recruitment.
* Active hepatitis B and C infection (positive HBV sAg and HBV-DNA more than 1x10^3 copies/mL; HCV-RNA more than 1x10^3 copies/mL) .
* Positive HIV antibody.
* Previous or current co-occurrence of other malignancies (except for effectively controlled non-melanoma basal cell carcinoma of the skin, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment in the past 5 years) .
* Primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at the time of recruitment.
* Pregnant or lactating female subjects and those who do not want to take contraceptive measures.
* Drug abuse (non-medical use of narcotic drugs or psychotropic drugs) or drug dependence (sedative hypnotics, analgesics, anesthetics, excitants and psychotropic drugs, etc.).
* A history of mental disease or cognitive impairment.
* Other conditions that the investigator determined are not suitable for participation in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence rate | From date of treating with conditioning regimen until lymphoma relapse, the end of follow-up or the date of death from any cause, whichever came first, assessed up to 36 months.
  The rate of lymphoma relapse

SECONDARY OUTCOMES:
AEs | From date of treating with conditioning regimen until the end of follow-up or the date of death from any cause, whichever came first, , assessed up to 36 months.
  adverse effects
Time of neutrophil implantation | From date of the treatment with the conditioning regimen until the time of neutrophil implantation or date of death from any cause, whichever came first, assessed up to 36 months.
  On the first day of three consecutive days, the peripheral blood neutrophil count (ANC) was ≥0.5×10^9/L without blood transfusion.
Time of platelet implantation | From date of the treatment with the conditioning regimen until the time of platelet implantation or date of death from any cause, whichever came first, assessed up to 36 months.
  On the first day of three consecutive days, the peripheral blood platelet count (PLT) was ≥20×10^9/L without blood transfusion.
OS | From date of treating with conditioning regimen until the end of follow-up or the date of death from any cause, whichever came first, , assessed up to 36 months.
  Overall survival
PFS | From date of treating with conditioning regimen until the end of follow-up or the date of death from any cause, whichever came first, , assessed up to 36 months.
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Pengcheng He, MD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China